CLINICAL TRIAL: NCT00618865
Title: Omega-3 Polyunsaturated Fatty Acids in Women With Major Depressive Disorders During Pregnancy
Brief Title: Omega-3 Fatty Acids for Major Depressive Disorder During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Kuan-Pin Su, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSC 93-2320-B-039-001
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2008-02

CONDITIONS: Depressive Disorder
Keywords: Omega-3 Fatty Acids; Major Depressive Disorder; Pregnancy; Women during pregnancy and after childbirth are more vulnerable to psychiatric disorders; Pharmacotherapy for depression during pregnancy is a clinical dilemma.; Omega-3 polyunsaturated fatty acids (PUFAs) might be a promising alternative of treatment for pregnant women with depression.
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): omega-3 fatty acid with 2.2 g of eicosapentanoic acid (EPA) and 1.2 g of docosahexanoic acid (DHA)
  Interventions: Dietary Supplement: Omega-3 fatty acids
- 2 (Placebo Comparator): Placebo (olive oil ethyl esters)
  Interventions: Dietary Supplement: Omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids

SUMMARY:
Whether high-dose omega-3 fatty acids supplement would be an effective treatment in patients with major depressive disorder during pregnancy and breast-feeding.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were pregnant women, aged 18 to 40 years, with major depressive disorder onset between their 16th week (second trimester) and 32nd week (third trimester) of gestation at the Department of Obstetrics.

Exclusion Criteria:

* Subjects were excluded with a DSM-IV diagnosis of bipolar disorders, psychotic disorders, substance abuse or dependence for at least 3 months, or any Axis-II diagnosis of borderline or antisocial personality disorder.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2004-06; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

REFERENCES:
- [Derived] Su KP, Huang SY, Chiu TH, Huang KC, Huang CL, Chang HC, Pariante CM. Omega-3 fatty acids for major depressive disorder during pregnancy: results from a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2008 Apr;69(4):644-51. doi: 10.4088/jcp.v69n0418. PMID 18370571